CLINICAL TRIAL: NCT00495417
Title: Randomized, Controlled, Parallel Group, Patient-blinded, Single-center Phase I Pilot Study to Assess Tolerability and Safety of Repeated s.c. Administration of a Single-dose of Affitope AD01 Applied With or Without Adjuvant to Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Tolerability and Safety of Subcutaneous Administration of Affitope AD01 in Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Affiris AG (Industry)
Responsible Party: Affiris GmbH
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Affiris 001; EUDRACT Number 2006-007063-90
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2009-09

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer; Morbus Alzheimer; Alzheimer Vaccine; Vaccine; AD; Aβ immunotherapy
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Biological: AFFITOPE AD01
- 2 (Active Comparator)
  Interventions: Biological: AFFITOPE AD01 adjuvanted

INTERVENTIONS:
Biological: AFFITOPE AD01 — s.c. injection
  Arms: 1
Biological: AFFITOPE AD01 adjuvanted — s.c. injection
  Arms: 2

SUMMARY:
The purpose of this study is to assess the tolerability and safety of repeated subcutaneous injection of a single dose of Affitope AD01 in patients with mild to moderate Alzheimer's Disease.

DETAILED DESCRIPTION:
Alzheimer's Disease (AD) is a devastating neurodegenerative disorder for which there is no cure.

Although the etiology of AD is not fully understood, recent research suggests that Aβ is central to the disease process. Consequently, approaches capable of removing Aβ from the brain, such as Aβ immunotherapy, are expected to possess disease-modifying potential. This view is supported by evidence gathered in mouse models of AD and studies involving AD patients.

Based on the view that active Aβ immunotherapy has disease-modifying potential both in animal models of AD and in patients, and on the knowledge gathered on the side-effects of Aβ-based immunotherapy encountered in humans, we designed a new generation of AD vaccines. Rather than using full length Aβ itself, we choose to use mimotopes of the N-terminal end of Aβ as the antigenic component of our vaccine (Mimotopes discovered by Affiris GmbH have been termed Affitopes). Mimotopes are peptides that functionally mimic the native antigenic epitope but do not show sequence identity to it. Thus, while being different from the original antigen, mimotopes are recognized by the same antibodies and, vice versa, are capable of inducing antibodies that cross-react with the original antigen itself. A major advantage offered by mimotopes is the lack of tolerance mechanisms that would prevent the induction of an immune response to it (as is the case with self peptides/proteins such as Aβ). To further increase the vaccine's safety profile, the length of the mimotope used was limited to preclude the elicitation of Aβ-specific T cells. Also, the mimotope used has been designed to generate antibodies directed exclusively to Aβ (i.e., they do not recognize parental APP itself). To provide helper epitopes for the generation of an antibody response, the mimotope is coupled to a carrier.

The trial is designed as a patient-blinded, single-center, randomized, controlled, parallel group, phase I clinical study of repeated once every 4 weeks administration by subcutaneous injection of Affitope AD01 alone or adsorbed to aluminum hydroxide in 24 patients with mild to moderate Alzheimer's Disease. In total, each patient will receive 4 immunizations. Patients will be randomized to receive Affitope AD01 alone or adsorbed to aluminum hydroxide. Each treatment group consists of 12 patients. For safety reasons, inclusion of patients will be done in a stepwise manner.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer's disease based on the NINCDS/ADRDA criteria.
* Assessing the severity of Alzheimer's disease of mild to moderate degree by the Mini Mental State Examination (MMSE 16-26)
* Hachinski Ischemia Scale ≤ 4.
* Magnetic Resonance Imaging scan (MRI) of brain consistent with diagnosis of AD.
* Informed consent capability (as determined by an independent neurologist)
* Written informed consent signed and dated by the patient or the patient's legal representative and the caregiver.
* Age >50 years.
* Availability of a partner/caregiver knowing the patient and being able to accompany the patient to the visits and being available for the telephone interviews.
* Adequate visual and auditory acuity to allow neuropsychological testing.
* Female patients of childbearing potential using a medically accepted contraceptive method.
* AD therapies on stable doses for at least 3 months prior to Visit 1 and during the entire trial period.
* Stable doses of all other medications for at least 30 days prior to Visit 1 if considered relevant by the investigator.

Exclusion Criteria:

* Pregnant women.
* Sexually active women of childbearing potential not using a medically accepted birth control method.
* Presence or history of allergy to components of the vaccine.
* Contraindication for MRI imaging.
* Operation (under general anaesthesia) within 3 months prior to study entry and scheduled elective operation during the whole study period.
* Participation in another clinical trial.
* History of questionable compliance to visit schedule; patients not expected to complete the clinical trial.
* Prior and/or current treatment with experimental immunotherapeutics including IVIG or vaccines for AD.
* Prior and/or current treatment with immunosuppressive drugs, concurrent treatment with beta-blockers.
* History and/or presence of autoimmune disease.
* Recent (≤3 years since last specific treatment) history of cancer (Exceptions: basal cell carcinoma, intraepithelial cervical neoplasia).
* Major psychiatric disorder (e.g. schizophrenia), if considered relevant by the investigator.
* Active infectious disease (e.g., Hepatitis B, C).
* Presence and/or history of Immunodeficiency (e.g., HIV).
* Significant neurological disease other than AD.
* Significant systemic illness.
* History of stroke or seizure.
* Change in dose of standard treatments for AD within 3 months prior to visit 1.
* Change in dose of other previous and current medications within the last 30 days prior to visit 1, if considered relevant by the investigator.
* Alcoholism or substance abuse within the past year (alcohol or drug intoxication).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Tolerability | One year

SECONDARY OUTCOMES:
Immunological and clinical efficacy (evaluated in explorative manner) | One year

CONTACTS AND LOCATIONS:
Overall Officials: Markus Müller, UnivProf.Dr., Principal Investigator — Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria